CLINICAL TRIAL: NCT04283006
Title: A Study of CD20/CD22 Targeted CAR T-cell Therapy for Relapsed or Refractory Lymphoid Malignancies
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: He Huang (Other)
Collaborators: Yake Biotechnology Ltd. (Industry)
Responsible Party: Sponsor-Investigator, He Huang, Clinical Professor, Zhejiang University
Organization: Zhejiang University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CD20/CD22-ZhejiangU
Record Dates: First submitted 2020-02-20; First posted 2020-02-25 (Actual); Last update posted 2020-08-21 (Actual); Status verified 2020-08

CONDITIONS: Relapsed and Refractory; Lymphoid Hematological Malignancies
Keywords: lymphoid hematological malignancies; CAR T-cell therapy; CD20/CD22
MeSH Terms: conditions — Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Administration of CD20/CD22 dual Targeted CAR T-cells (Experimental): A dose levels of 3-5*10E6/kg are administrated for each subject.
  Interventions: Drug: CD20/CD22 dual Targeted CAR T-cells

INTERVENTIONS:
Drug: CD20/CD22 dual Targeted CAR T-cells — Each subject receive CD20/CD22 dual Targeted CAR T-cells by intravenous infusion
  Other Names: CD20/CD22 dual Targeted CAR T-cells injection

SUMMARY:
A Study of CD20/CD22 Targeted CAR T-cell Therapy for Relapsed or Refractory Lymphoid Malignancies.

DETAILED DESCRIPTION:
Relapsed/refractory hematological malignancies has a short survival time and a high mortality rate. A number of clinical trials in China and at abroad have shown that CAR T-cells targeting CD19 have a high remission rate and limited adverse effects in the treatment of relapsed/refractory leukemia, which has great clinical application prospect. The New England Journal (NEJM) reported in 2010 and 2013 that the Carl June's team at the University of Pennsylvania used CAR T-cells against CD19 to treat B-cell malignancies successfully. On August 30, 2017, the US FDA first approved Novartis CAR T-cells for the treatment of acute lymphocytic leukemia. Our center has completed the treatment of 33 cases of acute lymphoblastic leukemia with CAR-T cells targeting CD19, with a complete remission rate of 90% and 10 cases of lymphoma treated with CAR T-cells. At present, the international clinical trials of CD20 / CD22 dual-target CAR T-cells in the treatment of relapsed/refractory lymphoid hematological malignancies have achieved impressive results, but the number of patients needs to be further verified.

Based on the results of prior studies and the lack of effective treatment options for relapsed/refractory hematological malignancies, we have applied for a clinical trial of CD20 / CD22 dual-target CAR T-cells to treat relapsed/refractory hematological malignancy.

This is a single arm, open-label, single-center study. Patients with CD20 and CD22-positive relapsed/refractory hematological malignancies have an estimated survival of 2 years. The purpose is to evaluate the safety and effectiveness of CD20 / CD22 dual-target CAR T-cell therapy through this clinical trial study, and to provide clinical basis and experience for CAR T-cell technology in the treatment of clinical malignant hematological diseases.

ELIGIBILITY:
Criteria:

Inclusion Criteria:

Inclusion criteria applicable to ALL only:

1. Male or female aged ≥ 3 and <70 years old;
2. Histologically confirmed diagnosis of CD19+ B-ALL per the US National Comprehensive Cancer Network (NCCN) Clinical Practice Guidelines for Acute Lymphoblastic Leukemia (2016.v1);
3. Relapsed or refractory CD19+ B-ALL (meeting one of the following conditions):

   1. CR not achieved after standardized chemotherapy;
   2. CR achieved following the first induction, but CR duration is ≤ 12 months;
   3. Ineffective after first or multiple remedial treatments;
   4. 2 or more recurrences;
4. The number of primordial cells (lymphoblast and prolymphocyte) in bone marrow is >5% (morphology) and/or >1% (Flow cytometry);
5. Philadelphia-chromosome-negative (Ph-) patients; or Philadelphia-chromosome- positive (Ph+) patients who cannot tolerate TKI treatments or do not respond to 2 TKI treatments;

Inclusion criteria applicable to NHL only:

1. Male or female aged ≥ 18 and <70 years old;
2. Histologically confirmed diagnosis per WHO Classification Criteria for Lymphocytic Tumors 2016, including DLBCL(NOS), follicular lymphoma, Chronic lymphoblastic leukemia/small lymphoblastic lymphoma transforms DLBCL, PMBCL and high grade B cell lymphoma;
3. Relapsed or refractory DLBCL (meeting one of the following conditions):

   1. No remission or recurrence after receiving second-line or above second-line chemotherapy;
   2. Primary drug resistance;
   3. Recurrence after autologous hematopoietic stem cell transplantation;
4. According to Lugano 2014, there should be at least one evaluable tumor lesion.

Applicable standards for ALL and NHL:

1. HLA antibody(-) or HLA antibody(+) and HLA donor specific antibody(DSA)(-);
2. total bilirubin ≤ 51umol/L, ALT and AST ≤ 3 times of upper limit of normal, creatinine ≤ 176.8umol/L;
3. Echocardiogram shows left ventricular ejection fraction (LVEF) ≥ 50%;
4. No active infection in the lungs, blood oxygen saturation by sucking air is ≥ 92%;
5. Estimated survival time ≥ 3 months;
6. ECOG performance status 0 to 2;
7. Patients or their legal guardians volunteer to participate in the study and sign the informed consent.

Exclusion Criteria:

1. patients with extramedullary lesions, except those with CNSL (CNS-1) under effective control (for ALL patients only);
2. Confirmed diagnosis of lymphoblastic crisis of chronic myeloid leukemia, Burkitt's leukemia/lymphoma per WHO Classification Criteria (for ALL patients only);
3. Patients with hereditary syndrome such as Fanconi anemia, Kostmann syndrome, Shwachman syndrome or any other known bone marrow failure syndrome (for ALL patients only);
4. Patients with intracranial extralateral lesions (cerebrospinal fluid tumor cells and/or intracranial lymphoma invasion shown by MRI) (for NHL patients only) ;
5. Extensive involvement of gastrointestinal lymphoma (for NHL patients only);
6. Radiotherapy, chemotherapy and monoclonal antibody within 1 week before screening;
7. Have a history of allergy to any of the components in the cell products;
8. Prior treatment with any CAR T cell product or other genetically-modified T cell therapies;
9. According to the New York heart association (NYHA) cardiac function classification criteria, Subjects with grade III or IV cardiac insufficiency;
10. Myocardial infarction, cardioangioplasty or stenting, unstable angina pectoris, or other severe cardiac diseases within 12 months of enrollment;
11. Severe primary or secondary hypertension of grade 3 or above (WHO Hypertension Guidelines, 1999);
12. Electrocardiogram shows prolonged QT interval, severe heart diseases such as severe arrhythmia in the past;
13. History of craniocerebral trauma, conscious disturbance, epilepsy, cerebrovascular ischemia, and cerebrovascular hemorrhagic diseases;
14. Patients with severe active infections (excluding simple urinary tract infection and bacterial pharyngitis).
15. Indwelling catheters in vivo (e.g. percutaneous nephrostomy, Foley catheter, bile duct catheter, or pleural/peritoneal/pericardial catheter). Ommaya storage, dedicated central venous access catheters such as Port-a-Cath or Hickman catheters are allowed;
16. History of other primary cancer, except for the following conditions:

    1. Cured non-melanoma after resection, such as basal cell carcinoma of the skin;
    2. Cervical cancer in situ, localized prostate cancer, ductal cancer in situ with disease-free survival ≥ 2 years after adequate treatment;
17. Patients with autoimmune diseases requiring treatment, patients with immunodeficiency or requiring immunosuppressive therapy;
18. Patients with graft-versus-host disease (GVHD);
19. Prior immunizations with live vaccine 4 weeks prior to screening;
20. History of alcoholism, drug abuse or mental illness;
21. If HBsAg positive at screening, HBV DNA copy number detected by PCR in patients with active hepatitis B > 1000 (if HBV DNA copy number≤1000, routine antiviral therapy is required after enrollment), as well as CMV, hepatitis C, syphilis infection;
22. Concurrent therapy with systemic steroids within 1 week prior to screening, except for the patients recently or currently receiving inhaled steroids;
23. Patients who have participated in any other clinical studies within 2 weeks prior to screening;
24. Pregnant and breast-feeding women and the subjects who are fertile and unable to take effective contraceptive measures (regardless of the gender);
25. Any situations that the investigator believes may increase the risk of patients or interfere with the results of study.

Ages: 3 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-05-23 (Actual); Primary Completion 2023-05-23 (Estimated); Study Completion 2028-05-23 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity (DLT) | Baseline up to 28 days after CD20/CD22 targeted CAR T-cells infusion
  Adverse events assessed according to NCI-CTCAE v5.0 criteria
Incidence of treatment-emergent adverse events (TEAEs) | Up to 2 years after CD20/CD22 targeted CAR T-cells infusion
  Incidence of treatment-emergent adverse events [Safety and Tolerability]

SECONDARY OUTCOMES:
B-cell acute lymphocytic leukemia (B-ALL), MRD negative overall response rate (MRD- ORR) | 3 months
  Assessment of MRD negative overall response rate (MRD- ORR) at 3 months after CD20/CD22 targeted CAR T-cells infusion
B-ALL, Event-free survival (EFS) | Month 6, 12, 18 and 24
  From the first infusion of CD20/CD22 targeted CAR T-cells to the occurrence of any event, including death, relapse or gene relapse, disease progression (any one occurs first), and the last visit
B-ALL, Overall response rate (ORR) | Month 6, 12, 18 and 24
  Assessment of ORR (ORR = CR + CRi ) at Month 6, 12, 18 and 24
B-ALL, Overall survival (OS) | Month 6, 12, 18 and 24
  From the first infusion of CD20/CD22 targeted CAR T-cells to death or the last visit
B cell non-hodgkin's lymphoma (B-NHL), Overall response rate (ORR) | weeks 4, 12, months 6, 12, 18 and 24
  Assessment of ORR (ORR = CR + PR ) per Lugano 2014 criteria
B-NHL, disease control rate (DCR) | weeks 12, months 6, 12, 18 and 24
  Assessment of DCR (DCR=CR+PR+SD) per Lugano 2014 criteria

CONTACTS AND LOCATIONS:
Locations (1):
- The First Hospital of Zhejiang Medical Colleage Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No